CLINICAL TRIAL: NCT04889677
Title: A Single Ascending Dose Study To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of ACH 0144471 In Healthy Volunteers
Brief Title: Study of a Single Dose of Danicopan in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ACH471-001
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: Danicopan; ALXN2040; ACH-0144471; Factor D Inhibitor; Pharmacokinetics; Pharmacodynamics; Ascending Dose
MeSH Terms: interventions — danicopan; rhoA GTP-Binding Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1: 200 mg (Experimental): All participants (fasted) received either 200 mg of danicopan as a single oral dose or dose-matched placebo.
  Interventions: Drug: Danicopan; Drug: Placebo
- Group 2: 600 mg (Experimental): All participants (fasted) received either 600 mg of danicopan as a single oral dose or dose-matched placebo.
  Interventions: Drug: Danicopan; Drug: Placebo
- Group 3: 1200 mg (Experimental): All participants (fasted) received either 1200 mg of danicopan as a single oral dose or dose-matched placebo.
  Interventions: Drug: Danicopan; Drug: Placebo
- Group 4: 2400 mg (Experimental): All participants (fasted) received either 2400 mg of danicopan administered as 2 single doses of 1200 mg each, 12 hours apart, or dose-matched placebo.
  Interventions: Drug: Danicopan; Drug: Placebo
- Group 5: 1200 mg (Experimental): All participants (fed) received either 1200 mg of danicopan as a single oral dose or dose-matched placebo.
  Interventions: Drug: Danicopan; Drug: Placebo

INTERVENTIONS:
Drug: Danicopan
  Other Names: ACH-0144471 (formerly); ALXN2040; ACH-4471; ACH4471; 4471
Drug: Placebo

SUMMARY:
This was a single ascending dose, randomized, double-blind study assessing the safety, tolerability, pharmacokinetics, and pharmacodynamics of danicopan in healthy participants. Four different doses (200 milligrams [mg], 600 mg, 1200 mg, 2400 mg) and dose-matched placebo were administered under fasted and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy defined as having no clinically relevant abnormalities identified by a detailed medical history, physical examination, blood pressure and pulse rate measurements, 12-lead electrocardiogram, and clinical laboratory tests.
* Body mass index of 18 to 30 kilograms (kg)/meter squared with a minimum body weight of 50 kg.

Exclusion Criteria:

* History or clinically relevant evidence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* Any condition possibly affecting drug absorption (for example, gastrectomy), cholecystectomy to be considered acceptable.
* Body temperature ≥ 38°Celcius on Day -1 or Day 1 Hour 0; history of febrile illness or other evidence of infection within 14 days prior to study drug administration.
* Current tobacco/nicotine users; consumption of any alcohol within 72 hours before study drug administration or a history of regular alcohol consumption exceeding 21 drinks/week within 6 months of Screening; positive urine drug screen at Screening or Day -1.
* Clinically significant laboratory abnormalities at either Screening or Day -1.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2016-06-21 (Actual); Study Completion 2016-06-21 (Actual)

PRIMARY OUTCOMES:
Incidence Of Serious Adverse Events, Grade 3 Or 4 Adverse Events (AEs), AEs Leading To Discontinuation, And Clinically Significant Laboratory Abnormalities And Electrocardiogram Abnormalities | Day 1 through Day 28

SECONDARY OUTCOMES:
Area Under The Plasma Concentration-time Curve Extrapolated To Infinity (AUC0-inf) Of Danicopan Under Both Fed And Fasted Conditions | Up to 144 hours postdose
Maximal Plasma Concentration (Cmax) Of Danicopan Under Both Fed And Fasted Conditions | Up to 144 hours postdose
Time To Reach The Maximal Plasma Concentration (Tmax) Of Danicopan Under Both Fed And Fasted Conditions | Up to 144 hours postdose
Relationship Between Alternative Pathway Inhibition And Danicopan Plasma Concentrations | Up to 144 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wiles JA, Galvan MD, Podos SD, Geffner M, Huang M. Discovery and Development of the Oral Complement Factor D Inhibitor Danicopan (ACH-4471). Curr Med Chem. 2020;27(25):4165-4180. doi: 10.2174/0929867326666191001130342. PMID 31573880